CLINICAL TRIAL: NCT01356069
Title: Sequential Brief Adlerian Psychodynamic Psychotherapy in Heavy Users of a Mental Health Service With Borderline Personality Disorder: a Two Years Follow-up Preliminary Randomized Study.
Brief Title: Efficacy of Time-limited Psychodynamic Psychotherapy and Informed Clinical Management in BPD High MHS Users
Acronym: HUMSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Prof. Secondo Fassino, University of Torino, Neurosciences Depatment
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUMHS-2004
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Heavy MHS Use; General Psychopathology; Working Alliance
Keywords: BPD; MHS; heavy users; sequential psychotherapy
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB-APP Psychotherapy (Experimental): Patients, who signed the informed consent, were randomly assigned to SB-APP in addition to TAU (n=18) or to TAU alone (n=17) groups. The SB-APP group received the usual treatment plus SB-APP (40 weekly sessions) for 10 or 11 months. At the term of the first year (T12) the TAU group continued with the TAU management with supportive weekly session whilst the SB-APP group was carried on with the psychiatric, nurse, educational management without any individual psychological support. The number of sessions performed by the two groups in the first year (T0-T12) was programmed to be almost the same to reduce the number of sessions bias comparing the specific quality of treatments.
  Interventions: Other: SB-APP
- TAU treatment (Active Comparator): This treatment consisted in a combination of medication, unstructured psychological support focused on socio-relational impairment and rehabilitative interventions provided by nurses and educators. The medication was administered according to the APA guidelines [18] for good clinical practice with regard to BPD.
  Interventions: Other: treatment as usual

INTERVENTIONS:
Other: SB-APP — SB-APP, derived from Brief-Adlerian Psychodynamic Psychotherapy (B-APP) is a time-limited (40 weekly sessions) psychodynamic psychotherapy based on Alfred Adler's theory and delivered in sequential and repeatable modules.
  SB-APP is focused specifically on four personality functioning levels (PFL). These are assessed by the therapists on the basis of symptoms, quality of interpersonal relationships, overall social behaviors, cognitive and emotional patterns, and defense mechanisms
  Arms: SB-APP Psychotherapy
Other: treatment as usual — This treatment consisted in a combination of medication, unstructured psychological support focused on socio-relational impairment and rehabilitative interventions provided by nurses and educators.
  Arms: TAU treatment

SUMMARY:
Subjects affected with severe Borderline Personality Disorder (BPD) are often heavy users of Mental Health Services (MHS). This study evaluates the efficacy of the addition of Sequential Brief Adlerian Psychodynamic Psychotherapy (SB-APP) to the treatment-as-usual (TAU) for BPD compared to the TAU alone for a naturalistic group of heavy MHS users with BPD. The efficacy was evaluated after at 6 time points along a two years of follow-up.

Thirty-five outpatients eligible for the study were randomly assigned to two treatment groups (TAU=17; SB-APP=18). The Clinical Global Impression (CGI) and the CGI-modified (CGI-M) for BPD, the Global Assessment of Functioning (GAF), the State-Trait Anger Expression Inventory (STAXI), and the Symptom Checklist-90 Revised (SCL-90-R) were administered at T1, T3, T6, T12, T18, and T24. At T12 also the Working Alliance Inventory-Short Form (WAI-S) was filled-in by participants and compared between groups. In the one-year follow-up the SB-APP group did not receive any individual psychological support. MHS was specifically trained in BPD treatment and had regular supervisions.

Scores of the CGI, GAF, and STAXI improved after 6 and 12 months, irrespective of treatment. SB-APP group displayed a better outcome for impulsivity, suicide attempts, chronic feelings of emptiness and disturbed relationships. The results displayed a good stabilization during follow-up year even after the interruption of psychotherapy in the SB-APP group.

Even though the TAU for BPD applied to heavy MSH users displayed some efficacy in reducing symptom expression and improving global functioning, the adjunct of a specific time-limited and focused psychotherapeutic treatment reached a better outcome. In particular the possibility of a focus on patients' personality functioning (SB-APP) with a specific psychotherapeutic approach seemed to be more effective than the general support to social impairment offered by the TAU approach.

ELIGIBILITY:
Inclusion criteria: (a) diagnosis of BPD according to DSM-IV-TR criteria; (b) age between 20 and 50 years; (c) heavy use of MHS during the year before the study - as defined below; and (h) signed informed consent.

Exclusion Criteria: (d) acute full-syndrome Axis I disorder requiring urgent inpatient treatment; (e) current Substance Dependence Disorder; (f) moderate to severe Mental Retardation; (g) previous treatment with structured psychotherapy;

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
MHS heavy use | 2 years
  requiring more than 6 emergency interventions per year

SECONDARY OUTCOMES:
psychopathological improvement | 2 years
  Clinical Global Impression (CGI) and the CGI-modified (CGI-M) for BPD, the Global Assessment of Functioning (GAF), the State-Trait Anger Expression Inventory (STAXI), and the Symptom Checklist-90 Revised (SCL-90-R) were administered at T1, T3, T6, T12, T18, and T24. At T12

CONTACTS AND LOCATIONS:
Overall Officials: Federico Amianto, MD, Principal Investigator — University of Torino; Andrea Ferrero, MD, Study Director — ASL TO-04 Chivasso (TO); Secondo Fassino, MD, Study Chair — University of Torino

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Amianto F, Ferrero A, Piero A, Cairo E, Rocca G, Simonelli B, Fassina S, Abbate-Daga G, Fassino S. Supervised team management, with or without structured psychotherapy, in heavy users of a mental health service with borderline personality disorder: a two-year follow-up preliminary randomized study. BMC Psychiatry. 2011 Nov 21;11:181. doi: 10.1186/1471-244X-11-181. PMID 22103890